CLINICAL TRIAL: NCT05975437
Title: Effectiveness of persoNalized Care After Treatment for Nonmetastasized Breast Cancer Based On Risk of Recurrence, Personal Needs and Risk on (Late) Health Effects: the NABOR Study
Brief Title: Effectiveness of Personalized Surveillance and Aftercare for Breast Cancer
Acronym: NABOR
Status: Enrolling by invitation | Type: Observational
Sponsor: Comprehensive Cancer Centre The Netherlands (Other)
Collaborators: University of Twente (Other); Dutch Breast Cancer Association (Unknown); Borstkanker Onderzoek Groep (Network); Netherlands Institute for Health Services Research (Unknown)
Responsible Party: Principal Investigator, Sabine Siesling, Senior researcher, full professor, Comprehensive Cancer Centre The Netherlands
Other Study IDs: 10330032010001
Record Dates: First submitted 2023-06-28; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer; Breast Cancer Female; Survivorship
Keywords: breast cancer; aftercare; surveillance; personalization; cost-effectiveness
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Care as usual: Participants who are included during care as usual, before the hospital's transition to personalized follow-up. Care as usual is organized as 'one-size fits all' and does not take individual differences in prognoses and needs into account. For the majority of hospitals follow-up includes annual mammography and physical examination combined with discussing of the results of the mammogram and sometimes also the patient's needs.
- Personalized care: Participants who are included after the hospital's transition to personalized follow-up. After this transition, personalized follow-up becomes the standard form of care for all patients, regardless of their participation in this study. Participants of this group receive personalized follow-up, which is based on individual prognoses and needs. Personalized follow-up will be provided by the use of personalized surveillance (PSP) and personalized aftercare plans (PAP).
  Interventions: Other: personalized surveillance plans (PSP) and personalized aftercare plans (PAP)

INTERVENTIONS:
Other: personalized surveillance plans (PSP) and personalized aftercare plans (PAP) — The PSP contains decisions on the surveillance trajectory based on individual risks and needs, assessed with the 'Breast Cancer Surveillance Decision Aid' including the INFLUENCE prediction tool. The PAP contains decisions on the aftercare trajectory based on individual needs and preferences and available care resources, which decision-making is supported by a patient decision aid.
  Groups: Personalized care

SUMMARY:
Surveillance and aftercare for curatively treated primary breast cancer patients is currently mostly 'one-size-fits-all', but can be personalized based on patients' risk of recurrence (depending on patient-, tumor- and treatment-related characteristics) and their personal needs and preferences. The use of personalized surveillance (PSP) and personalized aftercare plans (PAP) based on individual risks and needs might reduce unnecessary burden to the patient, increase quality of life and lower the costs of follow-up.

The NABOR study will examine the effectiveness of personalized follow-up care, consisting of personalized surveillance (PSP) and personalized aftercare plans (PAP) incorporating individual recurrence risks and personal needs of breast cancer patients. The main question it aims to answer is: 'what is the effectiveness of personalized surveillance (PSP) and aftercare plans (PAP), compared to current follow-up care, on cancer worry and self-rated overall quality of life (EQ-VAS)'. Also the effect of PSP and PAP on health-related quality of life (EQ-5D), societal participation, risk perception, patient satisfaction, patients' need for support, shared decision-making, health care costs and resource use, cost-effectiveness, and number and severity of the detected recurrences will be investigated. Next, the uptake and appreciation of the personalized plans and related factors (patient, caregiver, hospital and societal/financial) will be evaluated.

Patients participating in the study will have to fill in several questionnaires and give consent for requesting data from the Netherlands Cancer Registry and from their electronic health records (EHR).

The use of personalized surveillance (PSP) and personalized aftercare plans (PAP) will be implemented stepwise over a period of nine months in ten participating hospitals. To collect observations of both pre- and post-transition to PSP and PAP, each hospital will include patients during the nine months before and after its transition to personalized care.

In the future, the results of this project, i.e. the developed tools, can also be used for personalization of survivorship care for other cancer survivors. More broadly, all findings will be actively shared with interested healthcare professionals and other interested parties in the Netherlands.

DETAILED DESCRIPTION:
1. Treatment of subjects: personalized follow-up Personalized Surveillance Plan (PSP): Around the first surveillance mammogram (i.e. one year after end of treatment), the personalized surveillance plan (PSP) is generated by means of the PSP decision aid, called the 'Breast Cancer Surveillance Decision Aid' (16). This Aid incorporates the INFLUENCE tool 3.0, which is a sequel of the INFLUENCE tool 2.0 (15) and will be developed during this project. Compared to INFLUENCE 2.0, INFLUENCE 3.0 will additionally include patients treated with neoadjuvant therapy a broader population than INFLUENCE 2.0 (including patients treated with neoadjuvant therapy) and will include a more recent population in order to provide more contemporary risk estimates that are applicable in a broader population. During an outpatient clinic visit, around the first surveillance mammogram (i.e. approximately one year after the diagnosis), the INFLUENCE 3.0 prediction tool, as part of the PSP decision aid, is completed by the HCP (i.e. surgical oncologist or nurse specialist) and patient together by filling in data on patient, tumour and treatment characteristics. The estimated personal risk will be explained to the patient and summarized on a leaflet that also outlines the options possible for the patient (e.g. annual mammogram or less frequent, duration of follow-up, how to deliver the result from the mammogram). The patient receives a personal account with which she can, at home, complete the PSP decision aid that provides information about different surveillance options and a value clarification exercise to help the patient to get insight in her personal needs and preferences. This helps the patient to consider the pros and cons of the different options. A summary sheet based on patients' answers, combined with the result of the first surveillance mammogram, is used in the next consultation to make shared decisions on a personalized surveillance plan (PSP).

   Personalized Aftercare Plan (PAP): To support creation of this PAP, a patient decision aid (PtDA) will be used, which assesses patients' needs, offers information and provides a summary of patients' needs and preferences regarding the aftercare trajectory. The content of this PtDA will be developed in five cocreation sessions with a multidisciplinary team of researchers, patient representatives and care providers. First, needs assessment studies among patients and care providers will be conducted, which results serve as input for the content of the PtDA. This content will be critically revised by the team and rewritten to B1 language level (Common European Framework of Reference for Languages). Usability will be tested, consisting of think-aloud sessions with patients and interviews by telephone among health care professionals.

   During aftercare consultation(s) in the first year after the end of patients' treatment, the HCP (i.e. nurse or nurse specialist) will introduce the PtDA to the patient. Next, patients access the online PtDA to complete a needs assessment and receive information about possible effects of breast cancer, available options and choices that she has concerning her aftercare trajectory and available resources for help and support. Patients can weigh options and fill in preferences and considerations. Once patients have completed the PtDA, a summary sheet will automatically be created, containing an overview of patient-reported needs, preferences and considerations, which can be used as a base for final decision-making on the PAP in a consultation with their care provider. These decisions will compose the PAP, which will most likely include decisions on organisation of aftercare (e.g. further support or referrals, mode of contact, involved care providers) and signals to seek care for and contact details. Since patients' needs may vary over time, the care provider can introduce the PtDA multiple times during the aftercare trajectory. Also the PAP might be re-evaluated and adapted during the aftercare trajectory, depending on patients' needs and arranged contact frequencies.
2. Sample size calculation: The sample size was estimated using a user-written script for mITS designs in the Statistical Analysis System (SAS) software program. Since there are two primary parameters, a Bonferroni correction will be used to correct for multiple testing and therefore set the statistical significance level at alpha=0.025 (two sided). The effects the investigators wish to measure are a difference of 1.52 on the Cancer Worry Scale (CWS; range 6-24) and a difference of 4.8 on the EQ-VAS score (range 0-100), which is part of the EQ-5D. This decision is based on the aim to detect a small to moderate difference of 0.4 times the standard deviation, which was found to be around 3.8 for the CWS and 12 for the EQ-VAS score in previous studies. From a clinical point of view, a difference of 1.52 on the CWS is relevant for the purpose to estimate the effectiveness of personalized follow-up: even a small decrease in cancer worry can lead to improved quality of life. A difference of 4.8 on the VAS score is considered to be clinically relevant as well. A correlation is expected between the first two measurements within one hospital of 80%, and this correlation is expected to drop to 50% when comparing the first with the last measurement. In addition, an intraclass correlation coefficient of 0.15 is assumed. Taken 25% loss-to-follow up into consideration, each hospital will have to include four patients per period of three weeks in order to detect a difference of 1.52 on the CWS and 4.8 on the VAS score with 84%. The total inclusion time per hospital is 26 periods (78 weeks, or approximately 18 months), which amounts to a number of 104 patients per hospital and a study population of N=1,040.
3. Statistical analyses: An overview of the demographic and clinical characteristics will be provided using descriptive statistics. Continuous data will be expressed as a mean with the standard deviation (SD), or the Interquartile range (IQR) where appropriate. Categorical data will be expressed as frequencies (%). All questionnaires will be analysed in accordance with their corresponding manual. Self-composed questions (i.e. perceived risk of recurrence, adjusted questions from the CQ-Breast Index, demographics) will be analysed per item.

   To assess the effectiveness of personalized surveillance and aftercare, all outcome parameters will be compared between the current-care and personalized-care groups. Time series patterns will be visualized pre- and post-personalization to assess possible change in pattern after implementation of the personalization, for each hospital separately and combined. In this way the investigators can identify any underlying trends, seasonal patterns and outliers.

   To test the change in level and slope associated with the personalization and to control for other (confounding and overall trend) effects, segmented regression analyses will be used in which piecewise regression lines are fitted to each segment of time series, allowing each segment to exhibit different trends. To correct for correlation between repeated measurements residual plots against time will be visually examined, which can additionally be statistically tested using the Durbin-Watson statistic. Autocorrelation will consequently be adjusted for by including the autocorrelation parameter in the segmented regression model. Intention-to-treat analyses are done to estimate the effectiveness of personalized follow-up on the outcomes of the questionnaires. The Bonferroni correction will be used to adjust for multiple testing.

   Patients included during the transition phase will be analysed as receiving current care or personalized care dependent on whether PSP and PAP was applied. Sensitivity analyses will be performed with and without the patients included during the transition period, since there may be differences between care provided during and after the transition phase.

   In case of missing data, the investigators will record the percentage of drop-out and missing at each follow-up timepoint. If necessary, multiple imputation (if the assumptions for this technique are met) will be performed to ensure accurate analysis. Thereafter, meta-analyses will be performed to evaluate the average intervention effect per patient group across all hospitals and the overall effect across all patient groups and hospitals.

   A cost-effectiveness and cost-utility analysis will be performed comparing costs and effects of "personalized follow-up care" versus "usual care", using a two-year (study-based; based on data from the current study) and lifetime (model-based; based on the study and extrapolations by means of data from literature) time horizon. Information will be derived on the impact on personalized follow-up care on cancer worries, QoL, healthcare costs and (shift in) resources.

   Direct healthcare costs based on activities extracted from the EHRs (e.g. number of mammograms, consultations) will be multiplied by costs described in 'Benchmark costs from the Netherlands' or from the 'Nederlandse Zorgautoriteit' (NZa). For the costs of the interventions (decision support tools), an activity-based costing method will be performed for development, use and maintenance of the decision support platforms. Indirect costs that will be taken into consideration are healthcare consumption outside the hospital and health-related productivity losses. Productivity losses will be calculated by means of the Friction cost method, according to the International Society of Pharmaco-economical Organization and Research (ISPOR) guidelines.

   The cost-effectiveness will be expressed in incremental costs per patient with a clinically relevant improvement on the CWS as primary outcome of the NABOR study. The cost-utility will be expressed in incremental costs per quality adjusted life years (QALYs) gained, obtained from the EQ-5D-5L (including the VAS). Long term consequences will be based on both the study results and literature to extrapolate the patient outcomes for a lifelong time horizon.

   The cost-effectiveness analysis will be performed according to the guidelines for economic evaluations of the Dutch Zorginstituut (ZIN).
4. Handling of data

Data sources for our study:

* NCR (Netherlands Cancer Registry): data (e.g. patient-, tumor- and treatment-related characteristics) are already gathered and part of the general data collection of the NCR
* Additional patient data from the EHR: collected during the project
* PROFILES: a data registry collecting answers on questionnaires during the project Handling of data: For obtaining the data form the NCR, additional patient data from the EHR and answers on questionnaires through PROFILES, the study participants will provide Informed Consent. Registration will be done by the PROFILES registry. In order to send questionnaires to participants, participants will be asked permission for registration of their name and email-address or postal address in the PROFILES registry. In order to combine answers on questionnaires with data from NCR and the EHR later on, the PROFILES registry also needs their patient number and date of birth. Participants will also be asked permission for registration of their patient number and date of birth in the PROFILES registry. After the patient signs Informed Consent, the HCP will register the patient in PROFILES. HCPs can obtain the personal data and sequence number in the PROFILES registry, but have no access to the answers on questionnaires.

Accessibility of data: All the collected data is patient data, this cannot be made publicly available. Data from the NCR and additional EHR data can be requested, a local privacy committee evaluates requests. PROFILES data (i.e. answers on questionnaires) can be requested as well, and linked to NCR data if needed.

ELIGIBILITY:
Inclusion Criteria:

* female,
* aged 40 years or older (because of higher risk on recurrence),
* facing the decision for the organization of post-treatment surveillance and aftercare,
* being curatively treated including breast surgery, for invasive non-metastasized breast cancer
* able to understand the Dutch language in speech and writing.

Exclusion Criteria:

* bilateral breast cancers,
* BRCA1/2 or CHEK2 carriers,
* having an indication for MRI
* participation in another study that requires fixed scheduled follow-up consultations and/or imaging.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All new female patients who were curatively treated for non-metastasized primary breast cancer and start follow-up care in the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1040 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2027-03-06 (Estimated); Study Completion 2027-03-06 (Estimated)

PRIMARY OUTCOMES:
Change in cancer worry | 3 timepoints within 2 years: at T1 (1 year after end of treatment), T3 (2 years after end of treatment) and T5 (3 years after end of treatment)
  Cancer Worry Scale (CWS); Range 6-24, higher scores indicate greater worrying
Change in overall quality of life | 3 timepoints within 2 years: at T1 (1 year after end of treatment), T3 (2 years after end of treatment) and T5 (3 years after end of treatment)
  EQ-VAS (visual analogue scale of the EQ-5D); Range 0-100, higher scores indicate greater health-related quality of life

SECONDARY OUTCOMES:
Change in health-related quality of life on five domains | 3 timepoints within 2 years: at T1 (1 year after end of treatment), T3 (2 years after end of treatment) and T5 (3 years after end of treatment)
  Quality of life questionnaire (EQ-5D-5L); higher score indicate better quality of life
Change in health-related quality of life, concerning mental and physical domains | 3 timepoints within 2 years: at T1 (1 year after end of treatment), T3 (2 years after end of treatment) and T5 (3 years after end of treatment)
  Short-Form health index (SF-12); higher scores indicate greater quality of life
Change in health-related quality of life, concerning physical symptoms | 3 timepoints within 2 years: at T1 (1 year after end of treatment), T3 (2 years after end of treatment) and T5 (3 years after end of treatment)
  European Organization for Research and Treatment for Cancer Quality of Life Questionnaire (EORTC-QLQ-C30); higher scores indicate better health-related quality of life
Work productivity | 5 timepoints within 2 years: at T1 (1 year after end of treatment), T2 (1,5 years after end of treatment), T3 (2 years after end of treatment), T4 (2,5 years after end of treatment) and T5 (3 years after end of treatment)
  iMTA Productivity Cost Questionnaire (iPCQ); measures absence from work, reduced productivity while at work and productivity losses related to unpaid work
Healthcare consumption | 5 timepoints within 2 years: at T1 (1 year after end of treatment), T2 (1,5 years after end of treatment), T3 (2 years after end of treatment), T4 (2,5 years after end of treatment) and T5 (3 years after end of treatment)
  iMTA Medical Consumption Questionnaire (iMCQ); measures frequency of visits to health care practitioners outside the hospital and the extent to which others needed to join the patient in going to these visits, and the use of home care and medication
Risk perception | 3 timepoints within 2 years: at T1 (1 year after end of treatment), T3 (2 years after end of treatment) and T5 (3 years after end of treatment)
  Self-composed questionnaire on perceived risk of recurrence, measuring perceived absolute and comparative risk, perceived comparative risk and perceived course of the risk over time
Shared decision-making | 1 timepoint within 2 years: at T1 (1 year after end of treatment)
  Shared Decision-Making Questionnaire (SDM-Q-9); range 0-45, higher scores indicate a greater level of perceived involvement in decision-making
Patients' role in decision-making | 1 timepoint within 2 years: at T1 (1 year after end of treatment)
  Control Preference Scale (CPS); assesses the patient's preferred and perceived degree of control when decisions about treatment are being made. Higher scores indicate a preference for higher level of control in decision making
Patient satisfaction | 3 timepoints within 2 years: at T1 (1 year after end of treatment), T3 (2 years after end of treatment) and T5 (3 years after end of treatment)
  Consumer Quality breast care (CQ-breast index); higher scores indicate a greater satisfaction
Societal participation | 3 timepoints within 2 years: at T1 (1 year after end of treatment), T3 (2 years after end of treatment) and T5 (3 years after end of treatment)
  Lubben Social Network Scale (LSNS); higher scores indicate greater social engagement
Need for support for fear of cancer recurrence | 3 timepoints within 2 years: at T1 (1 year after end of treatment), T3 (2 years after end of treatment) and T5 (3 years after end of treatment)
  Questionnaire as composed by Luigjes-Huizer and colleagues, assesses the need for and experiences with support for fear of cancer recurrence

OTHER OUTCOMES:
Health literacy | 1 timepoint within 2 years: at T1 (1 year after end of treatment)
  Set of Brief Screening Questions (SBSQ); An average score of ≤2 indicates inadequate health literacy, and a score >2 indicates adequate health literacy
Mental adjustment to cancer | 1 timepoint within 2 years: at T1 (1 year after end of treatment)
  Mental Adjustment to Cancer scale (MAC); higher scores represent greater severity of the behaviors in the patient's struggle with cancer
Clinical characteristics, obtained from patients' Electronic Health Records | up to 2 years
  Performance of imaging (i.e. conclusion of imaging, breast density) and pathology (i.e. type of biopsies, cytology, histology), detected recurrences
Provided aftercare and surveillance; obtained from patients' Electronic Health Records | up to 2 years
  Information on frequency and reason of breast cancer-related hospital visits. This also includes (if applicable): information on decisions made about aftercare and surveillance, whether prediciton models or decision aids are used and whether aftercare and survaillance plans are personalized.
Tumor and treatment characteristics obtained from the Netherlands Cancer Registry | up to 2 years
  Tumour- and treatment-related characteristics, like tumour and nodal stage, differentiation grade, receptor status, radiotherapy, systemic therapy, targeted therapy, possible recurrences.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Siesling, Principal Investigator — Comprehensive Cancer Center of The Netherlands
Locations (10):
- Netherlands (10):
  - Gelre Ziekenhuizen, Apeldoorn, Gelderland
  - Rijnstate, Arnhem, Gelderland
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch, North Brabant
  - Bernhoven Ziekenhuis, Uden, North Brabant
  - Noordwest Ziekenhuisgroep, Alkmaar, North Holland
  - Ziekenhuisgroep Twente, Hengelo, Overijssel
  - Isala Klinieken, Zwolle, Overijssel
  - Albert Schweitzer Ziekenhuis, Dordrecht, South Holland
  - Alrijne Ziekenhuis, Leiderdorp, South Holland
  - Haaglanden Medisch Centrum, The Hague, South Holland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Luigjes-Huizer YL, van der Lee ML, Richel C, Masselink RA, de Wit NJ, Helsper CW. Patient-reported needs for coping with worry or fear about cancer recurrence and the extent to which they are being met: a survey study. J Cancer Surviv. 2024 Jun;18(3):791-799. doi: 10.1007/s11764-022-01326-5. Epub 2022 Dec 30. PMID 36585574
- [Derived] Klaassen-Dekker A, Drossaert CHC, Van Maaren MC, Van Leeuwen-Stok AE, Retel VP, Korevaar JC, Siesling S; NABOR project group. Personalized surveillance and aftercare for non-metastasized breast cancer: the NABOR study protocol of a multiple interrupted time series design. BMC Cancer. 2023 Nov 14;23(1):1112. doi: 10.1186/s12885-023-11504-y. PMID 37964214